CLINICAL TRIAL: NCT05460247
Title: The Effect of Protein Sources on Urinary Stone Risk
Brief Title: Protein Sources Urinary Stone Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Proteinsourcesv1
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Kidney Stone Prevention
Keywords: Nephrolithiasis; Kidney stones; Protein
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi | interventions — Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pea protein diet (Experimental)
  Interventions: Dietary Supplement: Protein
- Whey protein diet (Experimental)
  Interventions: Dietary Supplement: Protein
- Soy protein (Experimental)
  Interventions: Dietary Supplement: Protein
- Rice protein (Experimental)
  Interventions: Dietary Supplement: Protein

INTERVENTIONS:
Dietary Supplement: Protein — Participants will receive a diet supplemented by the above protein

SUMMARY:
Prior studies have shown that the source of dietary protein can have a significant impact on urinary stone risk. However, whey and plant protein isolates have not been compared. This is an important distinction as protein supplements fortified foods are increasingly popular. Herein, we seek to investigate the effect of different protein supplements, in an otherwise identical diet, on urinary stone risk.

DETAILED DESCRIPTION:
Each participant will receive a pre-made diet for 5 days at a time, for a total of 4 cycles. Previous studies have shown urine values reach a constant within the first 3 days. Diet will be a constant baseline diet representative of a standard Mediterranean diet. Participants will receive this diet to eat at home for 5 days with a supplemental protein shake at each meal (3 times a day). Participants will be required to drink 2.5-3 liters of fluid daily. Caffeine may be ingested as caffeine pills. Excessive exercise will be discouraged during the treatment phase.

Diet will remain constant with respect to protein quantity and all other ingredients and will only change protein isolate source in supplemental protein shake.

On days 4 and 5 of the diet, participants will be asked to collect two consecutive 24-hour urines. Between each 5-day diet phase, a flexible washout period will be allowed in which participants may eat a self-selected diet to take a break from standardized meals. Participants may resume the next phase diet on a day which is convenient for planned 24-hour urine collection at the end of that phase. The break period is to last no longer than 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to complete the study
2. Healthy with no personal or family history of kidney stones

Exclusion Criteria:

1. Allergy to any protein isolates or menu items used in the study
2. History of calcium oxalate, cysteine, uric acid, or infection stones
3. Disorders of absorption: Celiac disease, Irritable Bowel Disease, chronic diarrhea, short gut
4. Systemic predisposition to stones: gout, congenital hyperuricemia, chronic diarrhea, insulin resistance, neoplastic disorders, hyperparathyroidism or renal tubular acidosis
5. Women who are currently pregnant or planning pregnancy within 2 years
6. Renal transplant recipient
7. Bedridden study participants (ECOG ≥ 3)
8. Uncorrected anatomical obstruction of the urinary tract
9. History of recurrent urinary tract infections (> 3 urinary tract infections/year proven by urine culture)
10. Exclusions due to medication use:

    1. Chronic use of lithium
    2. Long-term glucocorticoid use (> 7.5 mg prednisone daily for > 30 days prior to enrollment)
    3. Intake of narcotic medication on a daily basis for >30 days prior to enrollment
    4. Supplemental Vitamin C (> 1 g daily)
    5. Carbonic anhydrase inhibitors (acetazolamide, topiramate, zonisamide)
    6. high dose calcium supplementation (> 1,200 mg daily)
    7. Medications that may crystallize in the urine (guaifenesin, sulfonamides, triamterene, and the protease inhibitors indinavir and nelfinavir).
11. Non-English Speakers
12. History of Syndrome of Inappropriate Antidiuretic Hormone Secretion (SIADH)
13. Anatomical urologic abnormalities including ileal conduits, horseshoe kidney, megaureter or solitary kidney
14. Psychiatric conditions impairing compliance with the study
15. Vulnerable population (prisoner and/or cognitive impairment that the investigator feels will impact participant's ability to complete study activities)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Urinary stone risk | 3 months after beginning study
  24 hour urine panel and supersaturation for Calcium Oxalate and Uric Acid
Calcium Oxalate Inhibitor activity | 3-6 months after beginning study
  mmol of Oxalate added before spontaneous precipitation

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States